CLINICAL TRIAL: NCT06649682
Title: Safety, Tolerability, Imaging Characteristics, and Efficacy of 68Ga-NYM096/177Lu-NYM096 in the Treatment of Patients With Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: 68Ga-NYM096/177Lu-NYM096 in Metastatic ccRCC
Acronym: NYCRRLT
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: This trial has been suspended given the concerns of stomach adverse effect in the first dose of 177Lu-NYM096 treatment (one patient developed grade 3 radiation-induced gastritis).
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K6754
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging and therapy (Experimental): 68Ga-NYM096 PET/CT and 177Lu-NYM096
  Interventions: Drug: 68Ga-NYM096 PET/CT and 177Lu-NYM096

INTERVENTIONS:
Drug: 68Ga-NYM096 PET/CT and 177Lu-NYM096 — Patients recruited in this study will undergo 68Ga-NYM096 PET/CT to evaluate the expression of carbonic anhydrase 9. Those with high CA9 expression will undergo 177Lu-NYM096 treatment, starting from 50mCi and increasing to 100mCi, 150mCi, 200mCi at most using a 3+3 design.

SUMMARY:
This is a single-center, phase I study. Patients with metastatic clear cell renal cell carcinoma will be recruited in this study to (Phase A) evaluate using 68Ga-NYM096 PET/CT and to (Phase B) treat with 177Lu-NYM096.

The study will be conducted in two phases. The purpose is Phase A: to evaluate the safety, tolerability, and imaging characteristics of 68Ga-NYM096 Phase B: to evaluate the safety, tolerability, and recommended phase 2 dose of 177Lu-NYM096

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18y
2. Histologically or cytologically confirmed metastatic clear cell renal cell carcinoma
3. Progression after or cannot undergo standard therapy with tyrosine kinase inhibitor (TKI) treatment or TKI combined with immune checkpoint inhibitor treatment.
4. Presence of at least 1 non-irradiated tumor lesion detected at conventional imaging (computed tomography / magnetic resonance imaging (CT/MRI)) documented within 4 weeks prior to the 68Ga-NYM096 administration which should be measurable per response evaluation criteria in solid tumors (RECIST) v1.1.
5. ECOG= 0 or 1
6. Written informed consent.
7. For Phase B: 68Ga-NYM096 should meet the imaging inclusion criteria

Exclusion Criteria:

1. Any major surgery within 12 weeks before enrollment
2. Inability to stay in the scanner bed and keep still for the duration of the scan
3. Participants who have not had resolution of clinically significant toxic effects of prior systemic cancer therapy, surgery, or radiotherapy to Grade ≤1
4. EGFR no higher than 30ml/min*1.73m2
5. Inflammatory bowel disease
6. Phase A: TKI treatment within one week before 68Ga-NYM096 administration
7. Phase B: Participants who received any systemic antineoplastic therapy for the underlying disease and/or other investigational agents within a period which is ≤5 half-lives or ≤4 weeks (whichever is shorter).
8. Any previous CA IX-targeting treatment
9. Prior external beam radiation therapy (EBRT) to more than 25% of the bone marrow
10. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
(Phase A) The number to patients with treatment-emergent adverse event (TEAE) and serious adverse event (SAE) | From the start of 68Ga-NYM096 PET/CT to 1 week after the 68Ga-NYM096 PET/CT
(Phase B) The number of patients with dose-limiting toxicity (DLT) after the first treatment of 177Lu-NYM096 | From the start of 1st cycle of 177Lu-NYM096 treatment (each cycle is 8 weeks) to 8 weeks later.
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The dose administrated to the participants will start at 50mCi and increase to 100, 150, and 200mCi at most in differnt dosing groups. While the AEs will be monitered for 8 months (2 months after the 4th dose), the decision whether the dose can increase to the next higher group will be decided only upon the DLT between the 1st and 2nd cycle.

SECONDARY OUTCOMES:
(Phase A) Dosimetry of 68Ga-NYM096 | 1 month after the 68Ga-NYM096 PET/CT
(Phase A) Number of lesions detected by 68Ga-NYM096 PET/CT | 1 week after the 68Ga-NYM096 PET/CT
(Phase A) Tumor uptake of 68Ga-NYM096 | 1 week after the 68Ga-NYM096 PET/CT
(Phase A) Optimal imaging window of 68Ga-NYM096 PET/CT | 1 week after the 68Ga-NYM096 PET/CT
(Phase B) The number of patients with treatment-emergent adverse event (TEAE) and serious adverse event (SAE) after 177Lu-NYM096 | From the start of 1st cycle of 177Lu-NYM096 administration (each cycle is 8 weeks) to 8 months later (8 weeks after the 4th cycle of treatment).
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The administration of 177Lu-NYM096 costs about half an hour.
(Phase B) Dosimetry of 177Lu-NYM096 | 1 month after 177Lu-NYM096 treatment
(Phase B) Radioactive concentration of 177Lu-NYM096 in the blood at different time point after 177Lu-NYM096 administration | From the start of 1st cycle of 177Lu-NYM096 administration (each cycle is 8 weeks) to 168 hours later.
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The administration of 177Lu-NYM096 costs about half an hour.
(Phase B) Tumor uptake of 177Lu-NYM096 on post-therapy scan | 1 week after 177Lu-NYM096 administration
(Phase B) ORR (overall response rate) of 177Lu-NYM096 treatment | From the start of 1st cycle of 177Lu-NYM096 treatment (each cycle is 8 weeks) to 2 years later.
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The tumor reponse will be evaluated before each cycle during the treatment (roughly every 2 months) and every 3 months after the end of the 4th cycle until 2 years after treatment start or tumor progression.
(Phase B) DCR (disease control rate) of 177Lu-NYM096 treatment | From the start of 1st cycle of 177Lu-NYM096 treatment (each cycle is 8 weeks) to 2 years later.
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The tumor reponse will be evaluated before each cycle during the treatment (roughly every 2 months) and every 3 months after the end of the 4th cycle until 2 years after treatment start or tumor progression.
(Phase B) PFS (progression free survival) of 177Lu-NYM096 treatment | From the start of 1st cycle of 177Lu-NYM096 treatment (each cycle is 8 weeks) to 2 years later.
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The tumor reponse will be evaluated before each cycle during the treatment (roughly every 2 months) and every 3 months after the end of the 4th cycle until 2 years after treatment start or tumor progression.
(Phase B) DOR (duration of response) of 177Lu-NYM096 treatment | From the start of 1st cycle of 177Lu-NYM096 treatment (each cycle is 8 weeks) to 2 years later.
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The tumor reponse will be evaluated before each cycle during the treatment (roughly every 2 months) and every 3 months after the end of the 4th cycle until 2 years after treatment start or tumor progression.
(Phase B) OS (overall survival) of 177Lu-NYM096 treatment | From the start of 1st cycle of 177Lu-NYM096 treatment (each cycle is 8 weeks) to the date of first documented date of death from any cause, assessed up to 60 months.
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The tumor reponse will be evaluated before each cycle during the treatment (roughly every 2 months) and every 3 months after the end of the 4th cycle until 2 years after treatment start or tumor progression. The survival info will be followed every 6 months until all-caused death of participant, assessed up to 60 months.
(Phase B) PFS rate at 6 months of 177Lu-NYM096 treatment | 6 month after the start of 1st cycle of 177Lu-NYM096 treatment (each cycle is 8 weeks) .
  177Lu-NYM096 will be delivered to participants up to 4 cycles with the same dosing amount. Each cycle will start 8 +/- 1 weeks after the previous cycle. The tumor reponse will be evaluated before each cycle during the treatment (roughly every 2 months).

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Principal Investigator — Peking Uion Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol, ICF